CLINICAL TRIAL: NCT04182932
Title: A Randomized, Double-blind, Placebo-controlled, Phase 1 Clinical Trial to Investigate the Safety and Immunogenicity of CJ-40010 After Administration in Healthy Subjects
Brief Title: Safety and Immunogenicity of CJ-40010 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CJ_HFM_101
Record Dates: First submitted 2019-11-25; First posted 2019-12-02 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Hand, Foot and Mouth Disease
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- CJ-40010 EV71 A dose (Experimental): Inactivated EV71 vaccine(A dose) or placebo in 10 healthy adults (three doses, 28 days interval)
  Interventions: Biological: CJ-40010 EV71 vaccine A dose; Biological: Placebo
- CJ-40010 EV71 B dose (Experimental): Inactivated EV71 vaccine(B dose) or placebo in 10 healthy adults (three doses, 28 days interval)
  Interventions: Biological: CJ-40010 EV71 vaccine B dose; Biological: Placebo
- CJ-40010 CVA16 C dose (Experimental): Inactivated CVA16 vaccine(C dose) or placebo in 10 healthy adults (three doses, 28 days interval)
  Interventions: Biological: CJ-40010 CVA16 vaccine C dose; Biological: Placebo
- CJ-40010 CVA16 D dose (Experimental): Inactivated CVA16 vaccine(D dose) or placebo in 10 healthy adults (three doses, 28 days interval)
  Interventions: Biological: CJ-40010 CVA16 vaccine D dose; Biological: Placebo
- CJ-40010 Bivalent E dose (Experimental): Inactivated EV71/CVA16 vaccine(E dose) or placebo in 10 healthy adults (three doses, 28 days interval)
  Interventions: Biological: CJ-40010 Bivalent vaccine E dose; Biological: Placebo
- CJ-40010 Bivalent F dose (Experimental): Inactivated EV71/CVA16 vaccine(F dose) or placebo in 10 healthy adults (three doses, 28 days interval)
  Interventions: Biological: CJ-40010 Bivalent vaccine high dose; Biological: Placebo

INTERVENTIONS:
Biological: CJ-40010 EV71 vaccine A dose — Inactivated vaccine against EV71, three doses, 28 days interval
  Arms: CJ-40010 EV71 A dose
Biological: CJ-40010 EV71 vaccine B dose — Inactivated vaccine against EV71, three doses, 28 days interval
  Arms: CJ-40010 EV71 B dose
Biological: CJ-40010 CVA16 vaccine C dose — Inactivated vaccine against CVA16, three doses, 28 days interval
  Arms: CJ-40010 CVA16 C dose
Biological: CJ-40010 CVA16 vaccine D dose — Inactivated vaccine against CVA16, three doses, 28 days interval
  Arms: CJ-40010 CVA16 D dose
Biological: CJ-40010 Bivalent vaccine E dose — Inactivated vaccine against EV71/CVA16, three doses, 28 days interval
  Arms: CJ-40010 Bivalent E dose
Biological: CJ-40010 Bivalent vaccine high dose — Inactivated vaccine against EV71/CVA16, three doses, 28 days interval
  Arms: CJ-40010 Bivalent F dose
Biological: Placebo — Placebo, three doses, 28 days interval

SUMMARY:
This study aims to evaluate the safety and immunogenicity of CJ-40010 after administration in healthy subjects

DETAILED DESCRIPTION:
Enterovirus 71(EV71) and coxsackievirus A16(CVA16) are major causes of Hand-foot-and-mouth disease (HFMD) occurring in pediatric population. Although EV71 vaccine has been licensed in China, vaccine for CVA16-associated HFMD is currently not available anywhere. The purpose of this phase I study is to evaluate the safety and immunogenicity of EV71/CVA16 bivalent vaccine in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men and women aged ≥19 to <50 years at the time of screening tests
* Body mass index(BMI)* of ≥18.0 kg/m2 to ≤27.0 kg/m2, with body weight of ≥55.0 kg to ≤90.0 kg for men and ≥50.0 kg to ≤90.0 kg for women at the time of screening tests

  *BMI (kg/m2) = Body weight (kg) / {height (m)}2
* Determined by the investigator to be eligible for study participation based on the results of screening tests (medical examination by interview, physical examination, vital signs, ECG, and clinical laboratory tests) conducted within 4 weeks of the 1st IP administration
* Intact deltoid muscle* that allows administration of the investigational product

  *Those who have a wound, scar, tattoo, skin disorder or infection on the expected investigational product administration site (deltoid muscle) that can affect safety evaluation cannot enter the study
* Consent to use medically acceptable contraception* throughout the study

  *Medically acceptable contraception: Use of an intrauterine device with a demonstrated pregnancy failure rate, concurrent use of a barrier method (male or female) and spermicide, surgical contraception of the subject or partner (vasectomy, salpingectomy/tubal ligation, hysterectomy, bilateral oophorectomy)
* Negative finding from a pregnancy test (urine hCG) at the time of the screening visit, after using medically acceptable contraception prior to 30 days of screening for women of childbearing potential*

  *Women of childbearing potential: Women who have not passed 1 year after menopause or not surgically sterilized (hysterectomy, bilateral oophorectomy)
* Voluntary decision and provision of written consent on participation in this study

Exclusion Criteria:

* History of a hand-foot-mouth disease or history of a disease related with enterovirus(EV) infection such as herpangina, viral meningitis, encephalitis, acute hemorrhagic conjunctivitis or myocarditis within 3 months prior to the 1st IP administration
* Medical history of an anaphylactic or similar acute reaction to CJ-40010 or similar vaccine
* Febrile disease or infectious disease within 2 weeks prior to the 1st IP administration
* Whole blood donation within 2 months or apheresis within 1 month prior to the 1st IP administration
* Vaccination with other prevention vaccine within 2 months prior to the 1st IP administration
* Use of an immunomodulator or immunosuppressant* within 3 months prior to the 1st IP administration

  * e.g., Azathioprine, Cyclosporin, Interferon, G-CSF, Tacrolimus, Everolimus, Sirolimus
  * High dose corticosteroids (continuous use for 14 days or more at ≥20 mg/day for Prednisolone. However, use of inhaled, intranasal or topical corticosteroids is allowed irrespective of the administered dose).
* History of a Guillain Barre syndrome
* Excessive caffeine intake (>5 units/day) or continuous alcohol consumption (>21 units/week, 1 unit = 10 g of pure alcohol) or incapable of abstention from alcohol during the study
* Participation in other clinical trial within 6 months prior to the 1st IP administration
* Pregnant or breastfeeding women
* Clinically significant hepatic, renal, neurological, respiratory, endocrine, hematology and oncology, cardiovascular, urological or psychiatric disease or such history
* Positive serological finding (type B hepatitis test, type C hepatitis test, human immunodeficiency virus(HIV) test)
* History of drug abuse or positive finding from a urine screening test for an abusive drug
* Use or of any prescription medication or oriental medicine within 2 weeks or any over-the-counter(OTC) medication, health functional food or vitamin within 1 week prior to the 1st IP administration (however, those who administered an allowed drug as specified in the other exclusion criterion can enter the study) or expected use of such products
* Administration of a blood product or blood-derived agent within 3 months prior to the 1st IP administration
* Determined by the investigator to be ineligible for study participation due to other reason including clinical laboratory findings

Ages: 19 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events of CJ-40010 (Safety of CJ-40010) | Week 0 to Week 32
  - Frequency and severity of adverse events up to 32 weeks post first dose

SECONDARY OUTCOMES:
Immunogenicity of CJ-40010 : Anti-EV71 IgG titer | Week 0 to Week 32
  Serum EV71-specific IgG titers
Immunogenicity of CJ-40010 : Anti-CVA16 IgG titer | Week 0 to Week 32
  Serum CVA16-specific IgG titers
Immunogenicity of CJ-40010 : Geometric mean titer (GMT) of EV71 neutralizing antibody titers | Week 0 to Week 32
  Geometric mean titers based on neutralizing antibody titers. Measurement of fold-increase over baseline of neutralizing titers against EV71
Immunogenicity of CJ-40010 : GMT of CVA16 neutralizing antibody titers | Week 0 to Week 32
  Geometric mean titers based on neutralizing antibody titers. Measurement of fold-increase over baseline of neutralizing titers against CVA16

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, Principal Investigator — Seoul National University Hospital, Dept. of Clinical Pharmacology
Locations (1):
- Seoul National University Hospital, Clinical Trial Center, Seoul, South Korea